CLINICAL TRIAL: NCT07014475
Title: Efficacy of the Ranger Drug-Coated Balloon in Treating Below-the-Knee Lesions in Patients With Chronic Limb-Threatening Ischemia
Brief Title: Efficacy of the Ranger Drug-Coated Balloon in Treating BTK Lesions in Patients With CLTI
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chang Guangqi, Clinical Professor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: [2025]194
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Chronic Limb Threatening Ischemia
Keywords: chronic limb threatening ischemia; below the knee; drug-coated balloon
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DCB: Ranger drug-coated balloon group
  Interventions: Device: drug-coated balloon

INTERVENTIONS:
Device: drug-coated balloon — Drug-coated balloon was used during the index procedure.

SUMMARY:
This is a prospective, multicenter, observational study designed to evaluate the clinical outcomes of the Ranger™ SL paclitaxel-coated balloon, a type of drug-coated balloon (DCB), in the treatment of below-the-knee (BTK) lesions in patients with chronic limb-threatening ischemia (CLTI) in China. All enrolled patients will be followed for six months. Patients diagnosed with CLTI who undergo treatment with the Ranger DCB will be included in the study. The primary outcome is the incidence of major adverse events (MAEs).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, gender is not limited
2. The patient agreed to participate in the CEIBA study and signed the written informed consent
3. Diagnosis of chronic limb-threatening ischemia (Rutherford category 4-6)
4. Gangrene involving any part of the lower extremities or feet, with exclusion of patients who have:

   4.1 Pure venous ulcers 4.2 Pure traumatic wounds 4.3 Acute limb ischemia (symptoms present for 2 weeks or less) 4.4 Embolic disease 4.5 Non-atherosclerotic chronic lower extremity vascular diseases (e.g., vasculitis, Buerger's disease, radiation arteritis)
5. Outflow Tract Requirement: At least one direct or indirect, unobstructed outflow vessel in the submalleolar segment of the target limb planned for revascularization.
6. Lesion Type:

6.1 Unobstructed blood flow in the suprapopliteal access pathway (including inflow vessels that have been recanalized via staged or concurrent endovascular intervention or hybrid surgery).

6.2 Sub-knee stenotic lesions ≥ 5 cm in length with ≥ 70% diameter reduction. 6.3 Sub-knee occlusive lesions ≥ 1 cm in length. 6.4 Two separate lesions with a minimum 3 cm interval between them may be considered as a single lesion for study inclusion purposes.

Exclusion Criteria:

1. Presence of life-threatening diseases or comorbidities with an expected life expectancy of less than 1 year.
2. Concurrent participation in another interventional clinical trial requiring informed consent.
3. Diagnosis of Alzheimer's disease.
4. Hematologic disorders or known bleeding tendency.
5. Contraindications to antiplatelet or anticoagulant therapy.
6. Known allergy to contrast agents that cannot be managed with standard premedication (e.g., steroids).
7. Deficiency or dysfunction of protein C, protein S, or antithrombin III (ATIII).
8. New York Heart Association (NYHA) Class III or IV heart failure.
9. Pregnancy or lactation.
10. Prior suprapatellar or infrapatellar amputation of the target limb.
11. Presence of aneurysm, perforation, dissection, or other target vessel injury requiring intervention.
12. Presence of other comorbid conditions (unrelated to the index disease) that affect walking function.
13. History of cardiovascular events within the past 3 months, including nonfatal myocardial infarction, unstable angina, stable angina, nonfatal ischemic stroke, or hemorrhagic stroke.
14. Clinically significant liver or renal dysfunction, as determined by the investigator.
15. Any other condition that, in the opinion of the investigator, would interfere with study treatment or functional assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with below-the-knee (BTK) arterial lesions diagnosed with chronic limb-threatening ischemia (CLTI).
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Events (MAEs) | 1 month; 3 months; 6 months
  Composite of target lesion revascularization (TLR), target limb amputation, and all-cause mortality.

SECONDARY OUTCOMES:
Late Lumen Loss (LLL) | 1 month; 3 months; 6 months
  Late lumen loss at the target lesion, measured by Quantitative Vascular Angiography (QVA).
Postoperative Complications | During procedure and hospitalization (up to 7 days post-procedure)
  Incidence of procedure-related adverse events, including arterial dissection, perforation, rupture, distal embolization, acute thrombosis, pseudoaneurysm, and hematoma formation.
Quality of Life (QoL) | Baseline, 1 month; 3 months; 6 months
  Assessed using the VascuQol-25 questionnaire, scored on a scale from 1 (worst) to 7 (best). Quality-adjusted life years (QALYs) calculated by multiplying the health-related quality of life (HRQoL) index score by time spent in each health state.
Rutherford Classification | Baseline, 1 month; 3 months; 6 months
  Grading system (0-6) for evaluating the severity of peripheral artery disease (PAD) in the lower extremities.
Amputation-Free Survival (AFS) | 1 month; 3 months; 6 months
  Defined as survival without ipsilateral major amputation (above the ankle).
Limb Salvage | 1 month; 3 months; 6 months
  Freedom from major (above-ankle) amputation in the target limb.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Giudice C, Galloula A, Tiercelin C, Vilfaillot A, Alsac JM, Messas E, Dean CL, Larger E, Sapoval M. "Ranger BTK" a Prospective Single-Centre Cohort Study on a New Drug-Coated Balloon for Below the Knee Lesions in Patients with Critical Limb Ischemia. Cardiovasc Intervent Radiol. 2021 Jul;44(7):1017-1027. doi: 10.1007/s00270-021-02833-1. Epub 2021 May 4. PMID 33948700
- [Background] Soga Y, Iida O, Takahara M, Hirano K, Suzuki K, Kawasaki D, Miyashita Y, Tsuchiya T. Two-year life expectancy in patients with critical limb ischemia. JACC Cardiovasc Interv. 2014 Dec;7(12):1444-9. doi: 10.1016/j.jcin.2014.06.018. PMID 25523536
- [Background] Fowkes FG, Aboyans V, Fowkes FJ, McDermott MM, Sampson UK, Criqui MH. Peripheral artery disease: epidemiology and global perspectives. Nat Rev Cardiol. 2017 Mar;14(3):156-170. doi: 10.1038/nrcardio.2016.179. Epub 2016 Nov 17. PMID 27853158
- [Background] Scully RE, Arnaoutakis DJ, DeBord Smith A, Semel M, Nguyen LL. Estimated annual health care expenditures in individuals with peripheral arterial disease. J Vasc Surg. 2018 Feb;67(2):558-567. doi: 10.1016/j.jvs.2017.06.102. Epub 2017 Aug 25. PMID 28847660
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883